CLINICAL TRIAL: NCT00803166
Title: Bioequivalence of Three Halobetasol Propionate 0.05% Topical Creams
Brief Title: Randomized Study to Compare the Bioavailability of Three Halobetasol Propionate 0.05% Topical Creams
Status: Completed | Type: Observational
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 10316926
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Bioequivalence; Halobetasol Propionate
MeSH Terms: interventions — halobetasol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort Group 1: Subjects number 1 to 30
  Interventions: Drug: Halobetasol Propionate 0.05% Cream-Reference Product; Drug: Halobetasol Propionate 0.05% Cream-Test product 1; Drug: Halobetasol Propionate 0.05% Cream-Test Product 2
- Cohort Group 2: Subjects number 31 to 60
  Interventions: Drug: Halobetasol Propionate 0.05% Cream-Reference Product; Drug: Halobetasol Propionate 0.05% Cream-Test product 1; Drug: Halobetasol Propionate 0.05% Cream-Test Product 2

INTERVENTIONS:
Drug: Halobetasol Propionate 0.05% Cream-Reference Product — Small amount applied and evaluated over the course of three days
Drug: Halobetasol Propionate 0.05% Cream-Test product 1 — Small amount applied and evaluated over the course of three days
Drug: Halobetasol Propionate 0.05% Cream-Test Product 2 — Small amount applied and evaluated over the course of three days

SUMMARY:
The purpose of this study was to compare the relative vasoconstrictive effects of two test and one reference Halobetasol Propionate 0.05% Cream in healthy, female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non-tobacco using female subjects, 18 to 50 years of age
* Demonstrated blanching response to Reference Drug
* Body Mass Index (BMI) of 30 or less
* Good health as determined by lack of clinically significant abnormalities in medical history and clinical assessment, as judged by the Investigator
* Signed and dated informed consent form which meets all criteria of current FDA regulations

Exclusion Criteria:

* History of allergy to systemic or topical corticosteroids
* Presence of any skin condition or coloration that would interfere with the placement of test sites or the response or assessment of skin blanching
* Presence of medical condition requiring regular treatment with prescription drugs
* Drug or alcohol addiction requiring treatment in the past 12 months prior to dosing
* Use of any tobacco products in the 30 days prior to study dosing
* Use of any dermatological drug therapy on the flexor surface of the forearms within 30 days of dosing
* Receipt of any drugs as part of a research study within 30 days prior to study dosing
* Pregnant or lactating

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Community Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Vasoconstriction will be measured by the degree of skin blanching observed after treatment removal using a ChromaMeter | Over the course of three days